CLINICAL TRIAL: NCT05753969
Title: The Efficacy of "Mindtesion"is Measuring Attentional and the Startle Response Dysregulation in Children and Adolescents Suffering From Attention Deficit Disorder: With and Without Medication.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Geha Mental Health Center (Other)
Responsible Party: Principal Investigator, Iris Manor, Director of ADHD clinic, Dan Petach-Tiqva, Geha MHC, Clalit, Geha Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 01-20-GEH
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Attention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPH / AMPH Treatment (Experimental)
  Interventions: Device: MT1 Device
- Placebo (Placebo Comparator)
  Interventions: Device: MT1 Device

INTERVENTIONS:
Device: MT1 Device — Pre-and post-evaluation in MT1 device following stimulant treatment or placebo control
  Other Names: Mindtension Attention Algorithm

SUMMARY:
Double blind, placebo-controlled clinical study designed to evaluate Mindtension device and Protocol as a diagnostic tool in children diagnosed with ADHD

DETAILED DESCRIPTION:
Mindtension device measures the orbicularis muscle response to auditory stimuli, the device is backed up by an algorithm that calculate the several parameters of startle reflex such as the Paired-pulse inhibition (PPI), Habituation, and startle related indices.

Data collected by the device is used to evaluate the subject levels of attention, Hyperarousal and Impulsivity, by means of physiological EMG signals of the startle response.

Evaluating baseline differences in these parameters between ADHD and age matched healthy controls, and the possible improvement after psychostimulant medications.

ELIGIBILITY:
Inclusion Criteria:

(i) Children with ADHD according to DSM-5 criteria in a semi-structured interview by a senior psychiatrist.

(ii) Reaching 85 percent score on the ADHD-RS scale. (iii) Treated with a stimulant in the perceived optimal dosage.

Exclusion Criteria:

(i) autism spectrum disorder. (ii) chronic neurological disorders and chronic medical conditions (e.g., diabetes).

(iii) schizophrenia spectrum and other psychotic disorders. (iv) substance abuse (drugs or alcohol). (v) depression. (vi) hearing loss. (vii) lack of cooperation.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Mindtension EMG values | baseline and 1 hour post treatment
  startle reflex indices such as the Paired-pulse inhibition (PPI), Habituation, and startle response amplitude, eye-blink probability, amplitude coefficients, inter-trial variability
ADHD severity | Baseline
  ADHD-RS-IV questionnaire ADHD-RS-IV questionnaire
Impulsive dysregulation | Baseline
  Clinical Global Impression (CGI): Clinical Global Impression - Severity and Clinical Global Impression - Improvement (CGI-S, CGI-I, respectively)

SECONDARY OUTCOMES:
CBCL | Baseline
  A questionnaire filled by the parents to describe their children's behavioral and emotional problems, version CBCL/4 to 18
Changes in treatment | Baseline
  Tolerability, switching rate, changes in formulation is examined using information from electronic medical records three clinical follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- ADHD clinic, Dan Petach-Tiqva, Geha MHC, Clalit, Petah Tikva, Israel